CLINICAL TRIAL: NCT04862429
Title: Studio BoCCE: Ruolo Della Biopsia Sotto Guida CEM (Mammografia Con Mezzo di Contrasto) Nella Caratterizzazione Delle Calcificazioni Dubbie o Sospette (BIRADS R3, R4, R5) Non Associate a Masse.
Brief Title: Biopsy of Calcifications Under Contrast Enhancement Guide (BoCCE)
Acronym: BoCCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BoCCE
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Calcification
Keywords: biopsy; contrast enhanced mammography; calcification
MeSH Terms: conditions — Breast Neoplasms; Calcinosis

STUDY DESIGN:
Intervention Model Description: Test and treat randomized trial.
Who Masked: Outcomes Assessor
Masking Description: Pathology results will be blindly reviewed by external pathologists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contrast enhanced mammography guided biopsy (Experimental): Patients will be subjected to CESM; the two orthogonal mammographic projections, after intravenous administration of iodized contrast-enhancement (Omnipaque), will be performed.
  Surgical and medical treatments will be defined accordingly to the imaging and histological findings obtained with the experimental procedure.
  Interventions: Other: Contrast enhanced mammography guided biopsy (diagnostic procedure)
- mammography guided biopsy (Active Comparator): Patients will be subjected to stereotactic biopsy Mammotome as normal clinical practice.
  Surgical and medical treatments will be defined accordingly to the imaging and histological findings obtained with the standard procedure.
  Interventions: Other: Mammography guided biopsy (diagnostic procedure)

INTERVENTIONS:
Other: Contrast enhanced mammography guided biopsy (diagnostic procedure) — With visible contrast-enhancement, stereotactic biopsy will be performed under CESM guidance. After administration of an additional dose of iodized contrast-enhancement (Omnipaque), the insertion of the biopsy needle and the biopsy sampling will be targeted on the area of greatest enhancement in the context of calcifications. In the absence of contrast-enhancement, stereotactic biopsy Mammotome will be performed, using X-ray guidance. The insertion of the biopsy needle and biopsy will be targeted on the most suspicious calcification cluster or area. At the end of the procedure, a metal clip marker will be placed in the biopsy site; the placement will be verified with dual orthogonal mammography projection (as regular clinical practice).
  Other Names: Contrast enhanced spectral mammography guided biopsy
  Arms: Contrast enhanced mammography guided biopsy
Other: Mammography guided biopsy (diagnostic procedure) — For all lesions, stereotactic biopsy Mammotome will be performed, using X-ray guidance. The insertion of the biopsy needle and biopsy will be targeted on the most suspicious calcification cluster or area.
  At the end of the procedure, a metal clip marker will be placed in the biopsy site; the placement will be verified with dual orthogonal mammography projection (as regular clinical practice).
  Other Names: stereotactic biopsy
  Arms: mammography guided biopsy

SUMMARY:
Calcification clusters are 30-40% of recalls in mammographic screening, but have a low positive predictive value (~15%) for ductal cancer in situ (DCIS) or invasive cancer. These calcifications often need histological assessment with stereotaxic guided biopsy (Mammotome). With extended calcifications, choosing the best area to biopsy may be challenging.

The main objective of this 1:1 randomized controlled clinical trial is to compare the accuracy of the CESM guide (study arm with biopsy under CESM guidance) with the traditional Mammotome (control arm with biopsy under stereotactic guidance) in conducting the biopsy in the area of greatest malignancy/grade of the lesion, using as gold-standard the histological exam of the operating piece. Women recalled with indication to perform stereotactic biopsy for clusters of suspicious calcifications on mammography (BIRADS R3 or R4 or R5) not mass-associated will be included. Anticipated sample size is 100 women per arm.

DETAILED DESCRIPTION:
Rationale Suspicious calcifications requiring further assessment are about 30-40% of recalls in mammographic screening. Nevertheless these findings have low positive predictive value (~15%) for ductal cancer in situ (DCIS) or invasive cancer. However, these calcifications are more frequently sent to biopsy than other doubt or suspect findings, due the difficulty in resolving the suspect with ultrasounds or with other imaging techniques.

For their histological check a biopsy with stereotaxic guidance (Mammotome) should be performed; when calcifications appear in several distinct clusters or over extended area, it is difficult to choose the best area to biopsy.

CESM is a technique that fuses mammographic images able to capture the morphology of calcifications (not visible at MRI) and the enanchement due to metabolic cellular and tissue vascular changes (not visible at usual X-ray imaging). Contrast-enhanced mammography (CESM) allows the description of both morphology and distribution of calcifications and contrast enhancement (CE). In the identification of pathological calcifications, CESM showed 91% sensitivity, 84% specificity, 77% VPP and 93% VPN, providing additional information for cancer diagnosis and dimensional definition of the pathological area.

This technique has the potential to allow a better sampling when biopsing calcifications than standard stereotactic biopsy.

Main objective: to compare the accuracy of CESM guide vs. stereotactic Mammotome guide in conducting biopsy in the area of major malignancy/grade of lesion.

Secondary objectives:

Between the two arms:

* To compare the proportion of patients undergoing pre-operative imaging with contrast media administration (it is expected to be almost 100% in intervention arm, but also in control arm some women will require additional pre-surgery assessment with MRI);
* To compare the proportion of upgrading from DCIS G1/G2 in pre-operative biopsy to DCIS G3 in surgical specimen;
* To compare the sensitivity of biopsy in the diagnosis of microinvasive/invasive tumors (pathology on surgical specimen as reference);
* Waiting time between biopsy and surgery;

Within the CESM arm:

* To compare mammography and CESM in terms of accuracy in the definition of lesion size and multifocality;
* To evaluate the association between the intensity of enhancement at CESM and the grade of malignancy of the lesion at histological examination on surgical specimen.

Population Women recalled with indication to perform stereotactic biopsy for clusters of suspicious calcifications on mammography (BIRADS R3 or R4 or R5) not mass-associated will be included. Anticipated sample size is 100 women per arm; this sample size will give a 75% power to detect.

Neoadjuvant therapy cannot be considered as an exclusion criteria, since the referral would occur after the enrollment and randomization. However, since it is extremely rare that not-mass associated lesions characterized by calcifications would require neoadjuvant therapy, the investigators do not anticipate to include patients who will be referred to therapy before surgery. If this unlikely event happens, women referred to neaodjuvant therapy will be included in the study without contributing to the analyses on the main objective and secondary objectives involving a comparison with post-operative pathological assessment.

Intervention Potentially eligible women will be informed about the study by the investigator radiologist during the visit in which mammography results are communicated. Women who express the willingness to participate will be asked to sign the informed consent and randomized to one arm with a 1:1 ratio.

Women in the experimental arm will undergo CESM. If in the images contrast-enhancement is visible, stereotactic biopsy will be performed under CESM guidance. After administration of an additional dose of iodized contrast-enhancement (Omnipaque), the insertion of the biopsy needle and the biopsy sampling will be targeted on the area of greatest enhancement in the context of calcifications. In the absence of contrast-enhancement, stereotactic biopsy Mammotome will be performed, using X-ray guidance. The insertion of the biopsy needle and biopsy will be targeted on the most suspicious calcification cluster or area.

Women in the control arm will undergo stereotactic biopsy (with Mammotome), using X-ray guidance. The insertion of the biopsy needle and biopsy will be targeted on the most suspicious calcification cluster or area.

In both arms, at the end of the procedure, a metal clip marker will be placed in the biopsy site; the placement will be verified with dual orthogonal mammography projection (as regular clinical practice).

According to the test and treat study design, surgical and medical treatments will be defined accordingly to the imaging and histological findings obtained in the arm of allocation.

Outcomes The main outcome is the accuracy of biopsy in collecting material from the most significant area.

Other outcomes will allow to measure downstream consequences of the biopsy. Surgical specimen will be used as the reference standard.

Analyses Main analyses will be conducted according to intention to treat strategy. The outcomes accuracy of biopsy, proportion of patients undergoing pre-operative imaging with contrast (CSM or MRI), proportion of upgraded lesions, biopsy sensitivity for microinvasive/invasive tumors, waiting time between biopsy and surgery will be compared between arms.

The outcomes accuracy in the definition of lesion size and multifocality, and enhancement predictivity for grade malignancy will be analysed within the experimental arm comparing CESM and mammography images in the same woman (paired analysis).

ELIGIBILITY:
Inclusion Criteria:

* Women with clinical mammography and screening recalls with mammographic confirmation of clusters of suspicious calcifications (BIRADS R3 or R4 or R5) not mass-associated will be included, with indication to perform stereotactic biopsy, evaluated at the Breast Care Facility of AUSL-IRCCS in Reggio Emilia.

Exclusion Criteria:

* Women with contraindication to the administration of iodized contrast medium will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with positive mammography for calcifications without mass, requiring biopsy
Enrollment: 200 (Estimated)
Dates: Start 2021-07-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Distance in mm between the biopsy site and the area of greatest malignancy/grade in the operating piece. | Cross-sectional: the reference standard will be collected during surgery, usually 3 to 6 weeks after biopsy. In any case, it cannot be collected more than 6 months after biopsy.
  In patients sent to surgery, the main outcome will be determined on the operating piece by a single pathologist operating in blind, which will assess the type of lesion (B1-B5), invasiveness, grade, the extent of the lesion in mm, the percentage of invasive component, the distance in mm between the location of the biopsy and the area of greatest malignancy (DCIS G3 or invasive component).
  In patients not sent to surgery, the outcome will be determined by following the patients for a follow-up of at least 24 months, verifying if they have undergone surgery on that specific lesion during the follow-up (in particular if they have developed B5 lesions in situ or invasive in that location).

SECONDARY OUTCOMES:
Proportion of patients needing contrast imaging | Cross-sectional: the reference standard will be collected during surgery, usually 3 to 6 weeks after biopsy. In any case, it cannot be collected more than 6 months after biopsy.
  Proportion of patients undergoing exam of pre-operative imaging with contrast will be compared between the two arms (it is expected to be almost 100% in intervention arm, but also in control arm some women will require additional pre-surgery assessment with MRI)
Diagnosis upgrading | Cross-sectional: the reference standard will be collected during surgery, usually 3 to 6 weeks after biopsy. In any case, it cannot be collected more than 6 months after biopsy.
  Proportion of diagnosis upgraded from DCIS G1/G2 in pre-operative biopsy to DCIS G3 in surgical specimen in the two arms.
Biopsy sensitivity | The reference standard will be collected during surgery, usually 3 to 6 weeks after biopsy. Women not needing surgery (negative at biopsy) will be followed up for 24 months in orther to assess the presence of cancers.
  Sensitivity of biopsy in the diagnosis of microinvasive/invasive tumors (pathology on surgical specimen as reference)
Waiting time between biopsy and surgery | The outcome measure is the time from biopsy to first surgical intervention, usually this time is in the range of 3 to 6 weeks.
  Waiting time between biopsy and surgery compared in the two arms, measured only in women needing surgery.
Accuracy for lesion size | Cross-sectional: the reference standard will be collected during surgery, usually 3 to 6 weeks after biopsy. In any case, it cannot be collected more than 6 months after biopsy.
  Lesion size (in terms of maximum diameter) from imaging (mammography or CESM). The outcome will be compared in the same lesion (paired analysis) only for women in experimental arm. Pathological measure on surgical specimen will be the reference standard.
Accuracy for multifocality | Cross-sectional: the reference standard will be collected during surgery, usually 3 to 6 weeks after biopsy. In any case, it cannot be collected more than 6 months after biopsy.
  Presence of multifocality (dichotomous variable) from imaging (mammography or CESM). The outcome will be compared in the same lesion (paired analysis) only for women in experimental arm. Pathological judgement on surgical specimen will be the reference standard.
Association between enhancement and grade | Cross-sectional: the reference standard will be collected during surgery, usually 3 to 6 weeks after biopsy. In any case, it cannot be collected more than 6 months after biopsy.
  To evaluate the association between the intensity of enhancement at CESM and the grade of malignancy of the lesion at histological examination on surgical specimen. The association will be measured on the same lesions (paired analysis) including only women in the experimental arm.

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Pattacini, MD, Principal Investigator — AUSL-IRCCS Reggio Emilia
Locations (1):
- Azienda USL - IRCCS di Reggio Emilia, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: Yes
Completely anonimized IPD with main patients' characteristics, numerical test results (no images) and outcomes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Seven years since publication of the result about main outcome.
Access Criteria: A request to Area Vasta Emilia Nord Ethic Committee should be submitted.

REFERENCES:
- [Background] Narayan AK, Keating DM, Morris EA, Mango VL. Calling all calcifications: a retrospective case control study. Clin Imaging. 2019 Jan-Feb;53:151-154. doi: 10.1016/j.clinimag.2018.09.016. Epub 2018 Oct 5. PMID 30340079
- [Background] Si J, Guo R, Huang N, Xiu B, Zhang Q, Chi W, Wu J. Axillary evaluation is not warranted in patients preoperatively diagnosed with ductal carcinoma in situ by core needle biopsy. Cancer Med. 2019 Dec;8(18):7586-7593. doi: 10.1002/cam4.2623. Epub 2019 Oct 29. PMID 31660702
- [Background] Jakub JW, Murphy BL, Gonzalez AB, Conners AL, Henrichsen TL, Maimone S 4th, Keeney MG, McLaughlin SA, Pockaj BA, Chen B, Musonza T, Harmsen WS, Boughey JC, Hieken TJ, Habermann EB, Shah HN, Degnim AC. A Validated Nomogram to Predict Upstaging of Ductal Carcinoma in Situ to Invasive Disease. Ann Surg Oncol. 2017 Oct;24(10):2915-2924. doi: 10.1245/s10434-017-5927-y. Epub 2017 Aug 1. PMID 28766196
- [Background] Grimm LJ, Ryser MD, Partridge AH, Thompson AM, Thomas JS, Wesseling J, Hwang ES. Surgical Upstaging Rates for Vacuum Assisted Biopsy Proven DCIS: Implications for Active Surveillance Trials. Ann Surg Oncol. 2017 Nov;24(12):3534-3540. doi: 10.1245/s10434-017-6018-9. Epub 2017 Aug 9. PMID 28795370
- [Background] Cheung YC, Tsai HP, Lo YF, Ueng SH, Huang PC, Chen SC. Clinical utility of dual-energy contrast-enhanced spectral mammography for breast microcalcifications without associated mass: a preliminary analysis. Eur Radiol. 2016 Apr;26(4):1082-9. doi: 10.1007/s00330-015-3904-z. Epub 2015 Jul 10. PMID 26159872
- [Background] Iotti V, Ragazzi M, Besutti G, Marchesi V, Ravaioli S, Falco G, Coiro S, Bisagni A, Gasparini E, Giorgi Rossi P, Vacondio R, Pattacini P. Accuracy and Reproducibility of Contrast-Enhanced Mammography in the Assessment of Response to Neoadjuvant Chemotherapy in Breast Cancer Patients with Calcifications in the Tumor Bed. Diagnostics (Basel). 2021 Mar 4;11(3):435. doi: 10.3390/diagnostics11030435. PMID 33806306
- See also: European guidelines on breast cancer screening and diagnosis — http://healthcare-quality.jrc.ec.europa.eu/european-breast-cancer-guidelines